CLINICAL TRIAL: NCT06759051
Title: Targeted TDCS Intervention for Internet Gaming Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGD-tDCS
Record Dates: First submitted 2024-12-12; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Internet Gaming Disorder
Keywords: Internet gaming disorder; tDCS; IGD
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Active Intervention Group-Central parietal cortex (cathode) (Active Comparator): A 5*5cm square electrode sheet was placed in the subject's central parietal brain area (Pz electrode point) and a 5*5cm square electrode sheet was placed at the trapezius muscle at the base of the right side of the neck, where cathodic stimulation was given at the parietal lobe and anodic stimulation was given at the right trapezius muscle. Subjects will be intervened under a drug cue response task. The stimulation pattern of the true intervention is that the current level ramps up from 0 to 2mA in the first 10 seconds of stimulation onset, then maintains the 2mA level for a continuous stimulation period of 19 minutes and 40 seconds, and then decreases the current level from 2mA to 0mA in the last 10 seconds. the whole process lasts for 20 minutes.
  Interventions: Device: tDCS
- Sham Intervention Group-Central parietal cortex (cathode) (Sham Comparator): A 5*5cm square electrode sheet was placed in the subject's central parietal brain area (Pz electrode point) and a 5*5cm square electrode sheet was placed at the right trapezius muscle at the base of the neck, where cathodic stimulation was given at the parietal lobe and anodic stimulation at the right trapezius muscle. The whole process lasted 20 min. Subjects will be intervened under a drug cue response task. The sham intervention will be conducted in such a way that during the first 20 seconds of stimulation, the current will ramp up from 0mA to 2mA and then ramp down to 0mA, maintaining the current at 0mA for 19 minutes and 20 seconds, and then in the last 20 seconds, the current will ramp up from 0mA to 2mA and then ramp down to 0mA. The whole duration of the procedure will be the same as that of the real intervention.
  Interventions: Device: Sham (No Treatment)
- Active Intervention Group-Dorsolateral Prefrontal Cortex (anodic) (Active Comparator): A 5*5cm square electrode sheet will be placed in the subject's left DLPFC brain area (F3 electrode site) and a 5*5cm square electrode sheet will be placed at the right trapezius muscle at the base of the neck, where anodic polar stimulation will be given at the DLPFC and cathodic stimulation will be given at the trapezius muscle at the base of the neck on the right right side. Subjects will be intervened under a drug cue response task. The stimulation pattern of the true intervention is that the current level ramps up from 0 to 2mA in the first 10 seconds of stimulation onset, then maintains the 2mA level for a continuous stimulation period of 19 minutes and 40 seconds, and then decreases the current level from 2mA to 0mA in the last 10 seconds. the whole process lasts for 20 minutes.
  Interventions: Device: tDCS
- Sham Intervention Group-Dorsolateral Prefrontal Cortex (anodic) (Sham Comparator): A 5*5cm square electrode sheet will be placed in the subject's left DLPFC brain area (F3 electrode site) and a 5*5cm square electrode sheet will be placed at the right trapezius muscle at the base of the neck, where anodic polar stimulation will be given at the DLPFC and cathodic stimulation will be given at the trapezius muscle at the base of the neck on the right right side. Subjects will be intervened under a drug cue response task. The whole procedure lasts for 20 minutes. The sham intervention will be in the form of a current that ramps up from 0mA to 2mA and then ramps down to 0mA for the first 20 seconds of stimulation onset. after maintaining a current level of 0mA for 19 minutes and 20 seconds, the current will again ramp up from 0mA to 2mA for the last 20 seconds and then ramp down to 0mA.
  Interventions: Device: Sham (No Treatment)
- Active Intervention Group for EEG-tDCS (Active Comparator): The personalised EEG classifier model established through machine learning is used to identify the current game cue response EEG pattern state of the subject during intervention and perform tDCS intervention in real time. The real-time EEG data of the true intervention group was collected for 1 second at a time in real time, and then pre-processed, and feature extraction was performed on the real-time EEG data using the temporal clusters in the first part, and then inputted into the EEG classifier model mentioned above, which in turn calculated the similarity between the current state and the previous game cue response-evoked EEG pattern, i.e., whether or not it was currently in a high craving response state. Once in the high craving state and short-term tDCS intervention, the intervention site is the effective target site found above, and a short-term electrical stimulation intervention of 2 seconds and 2mA is given.
  Interventions: Device: tDCS
- Sham Intervention Group for EEG-tDCS (Sham Comparator): The EEG signal of the subject completing the game cue response task is first acquired, the signal is preprocessed, and then the time-domain voltage feature and the time-frequency domain energy feature of the EEG are obtained by comparing the game cue and the neutral cue condition, and the spatiotemporal clusters of the time-domain feature and the time-frequency domain feature under the above thresholds are obtained by the method based on the cluster statistic in the EEG analysis in the adjacent time window and the adjacent electrode position, respectively. Further, a personalised EEG classifier model is established by machine learning.
  The above model is used during intervention to identify the current EEG pattern state of the subject's game cue response and perform tDCS intervention in real time. The sham intervention group used the EEG data of the real intervention group for intervention triggering.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: tDCS — The stimulation pattern for the true intervention was that the current level ramped up from 0 to 2 mA for the first 10 seconds of stimulation, then maintained at 2 mA for 19 minutes and 40 seconds, and then ramped down from 2 mA to 0 mA for the last 10 seconds, all over a 20-minute period.
  Arms: Active Intervention Group for EEG-tDCS; Active Intervention Group-Central parietal cortex (cathode); Active Intervention Group-Dorsolateral Prefrontal Cortex (anodic)
Device: Sham (No Treatment) — In contrast to the active intervention, the sham intervention consisted of a current ramp from 0mA to 2mA for the first 20 seconds of stimulus onset, followed by a ramp down to 0mA. the current was maintained at 0mA for 19 minutes and 20 seconds, and then the current was ramped from 0mA to 2mA for the last 20 seconds, followed by a ramp down to 0mA. The entire procedure lasted the same as the active intervention, which lasted for 20 minutes.
  Arms: Sham Intervention Group for EEG-tDCS; Sham Intervention Group-Central parietal cortex (cathode); Sham Intervention Group-Dorsolateral Prefrontal Cortex (anodic)

SUMMARY:
The aim of this project is to compare the effects of the newly discovered parietal cortex (Pz electrode point) with the dorsolateral prefrontal cortex (F3 electrode point), which has been commonly used in previous studies, and to further develop a closed-loop intervention method of real-time tDCS under on-line electroencephalography (EEG-tDCS), so as to realise an individualised diagnosis and treatment for online game addicts.

This study is divided into two parts, the first part to explore the effectiveness of the new target, using a randomised group design, using tDCS intervention, the subject population is online game addicts, the sample size is about 120. Participants underwent baseline information collection on the first day of the experiment including: basic demographic information, assessment of internet addiction severity and craving; EEG collection in resting state as well as task state (Game Cue Response Task, Signal Stop Task, Iowa Gambling Task). The tDCS intervention under the game cue response task was conducted on the second and third days of the experiment, divided into four groups (the first and second groups were the true-false stimulation groups with the anode at the trapezius muscle at the base of the right neck and the cathode at the subject's central parietal cortex; and the third and fourth groups had the anode at the subject's left dorsolateral prefrontal cortex, and the cathode at the trapezius muscle at the base of the right neck), with 20 min of intervention each time and the Game craving level was assessed before and after the intervention. Resting-state and task-state (Game Cue Response Task, Signal Stop Task, Iowa Gambling Task) EEG acquisitions were performed at the end of the intervention.The second part of the EEG-tDCS closed-loop intervention was conducted, using a randomised group design with a sample size of about 60 subjects who are addicted to online games. On the first day of the experiment, baseline information was collected, and a personalised EEG classifier model was built for each subject based on the EEG signals of the game cue response task; on the second and third days of the experiment, EEG-tDCS closed-loop intervention was conducted, divided into true intervention and sham intervention groups, with the true intervention group identifying whether subjects were in an addictive state in real time under the game cue response task, and addictive states were identified by giving real-time short-time short-time short-time short-time short-time short-time short-time intervention at target locations. The real-time short-term tDCS intervention was given at the target location for a total duration of 20 minutes, and the level of game craving was assessed after the intervention; at the end of the intervention, the EEG was collected in the resting state and the task state (game cue response task, signal stopping task, and Iowa gambling task). The two-part experiment followed up subjects with weekly post-intervention versus one-month post-intervention gaming severity assessments, with resting-state and task-state (gaming cue-response task, signal-stopping task, Iowa gambling task) electroencephalogram acquisitions.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-30 years old; and
2. Familiar with and mainly play King's Honour;
3. IGDS9-SF score ≥ 32 points
4. Meets DSM-5 diagnostic criteria for online game addiction;
5. Played online games for at least 14 hours per week in the past 1 year;
6. signed an informed consent form to voluntarily participate in this trial.

Exclusion Criteria:

1. severe mental illness, neurological disorder or physical illness; and
2. History of substance abuse/dependence (including alcohol);
3. Contraindications to EEG acquisition;
4. Colour blindness, colour deficiency or other vision-related eye diseases affecting vision;
5. Pregnant and breastfeeding women, or women who are menstruating; and
6. Poor compliance: subjects who, in the opinion of the investigator, are unable to co-operate with the trial.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Craving Of Game (VAS) | "From enrollment to the end of treatment at 1 month"
  Subjects' thirst was indicated by scores on a questionnaire (VAS)，The range is 0-9, with 0 meaning that you don't want to play the game very much after looking at the picture, and 9 meaning that you want to play the game very much after looking at the picture.

SECONDARY OUTCOMES:
Craving Of Game (Questionnaire on Gaming Urge, Brief Version(QGU-B)) | "From enrollment to the end of treatment at 1 month"
  Subjects' thirst was indicated by scores on a questionnaire (QGU-B)，The QGU-B scale consists of 10 items, and the intensity of each item is indicated by a score from 1 to 7, with higher scores indicating a stronger urge to play.
Severity of game addiction (DSM-5) | "From enrollment to the end of treatment at 1 month"
  The severity of the subject's gaming addiction is indicated by the score on the questionnaire (DSM-5)，The DSM-5 scale consists of nine items, each of which has a "yes" or "no" choice, with a "yes" choice counting as one point and a "no" choice being indicated by a score from 1 to 7. "The higher the score, the more severe the online game use disorder.
Severity of game addiction (Internet Gaming Disorder Scale-Short-Form(IGD-S9)) | "From enrollment to the end of treatment at 1 month"
  The severity of the subject's gaming addiction is indicated by the score on the questionnaire (IGD-S9)，The IGD-S9 scale consists of nine items with scores ranging from 9 to 45, with higher scores indicating higher levels of addiction.
Electroencephalographic (EEG) index | "From enrollment to the end of treatment at 1 month"
  Brain waves of subjects in resting or task states, include P300 at Pz electrode, point；time frequency of P300 (alpha, theta, beta, delta).
Behavioural indicators under EEG tasks | "From enrollment to the end of treatment at 1 month"
  Under the Iowa Gambling task (IGT), participants were analyzed for the percentage of participants choosing each type of card (high-risk but high-reward, low-risk but low-reward), thus comparing their risky decision-making abilities; under the Signal Stopping task (SST), participants were analyzed for their stop-signal reaction time (SSRT), which is the amount of time it takes an individual to successfully inhibit a response that has been initiated, thus assessing response inhibition; and under the Monetary Incentive Delay task (MID), subjects were analyzed for five conditions (large win, large loss, small win, small loss, neutral ) reaction times and accuracy, assessing participants' expectations of rewards and punishments and outcome feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Dependence, Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No